CLINICAL TRIAL: NCT05513378
Title: A Randomized Controlled Trial Comparing In-line Ultrasound Guided Subclavian Vein Catheterization With or Without Needle Guide.
Brief Title: Ultrasound-guided Subclavian Vein Catheterisation With a Needle Guide
Acronym: ELUSIVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thomas Kander (Other)
Responsible Party: Sponsor-Investigator, Thomas Kander, Associate Professor and Sponsor Investigator, Region Skane
Organization: Region Skane (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: ELUSIVE
Record Dates: First submitted 2022-08-21; First posted 2022-08-24 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Complications; Catheter, Mechanical; Catheterization, Central Venous
Keywords: diagnostic imaging

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The researcher who will review the documented ultrasound movies and assess the secondary outcomes will be blinded. However, given the nature of the study neither the Care Provider or Investigators will be blinded for the group affiliation or the primary outcome
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- With Needle Guide (Experimental): A needle guide adapted to a micro-convex ultrasound probe will be used in ultrasound-guided catheterisation of the subclavian vein using the long-axis approach with an in-plane needling technique
  Interventions: Device: Needle guide
- Without Needle Guide (No Intervention): A micro-convex ultrasound probe without needle guide will be used in ultrasound-guided catheterisation of the subclavian vein using the long-axis approach with an in-plane needling technique

INTERVENTIONS:
Device: Needle guide — Please see the arm/group description
  Other Names: The Ultra-Pro II™ Needle Guide, model C8-5 Philips
  Arms: With Needle Guide

SUMMARY:
OBJECTIVES The primary objective is to compare if the addition of a needle guide can reduce the number of central venous catheter (CVC) insertions with >1 skin puncture in ultrasound-guided catheterization of the subclavian vein using the long-axis approach with an in-plane needling technique.

Secondary objectives include if this addition 1) decreases the frequency of mechanical complications (defined as bleeding, arterial puncture, arterial catheterization, nerve injury, pneumothorax), 2) increases the time when the needle is visible, 3) decreases the time until successful vessel punction, 4) decreases the number of needle redirections during the insertion, and 5) a comparison between the two groups regarding number of failed catheterizations.

DESIGN This is a prospective, randomised, controlled, parallel intervention study. Patients will be enrolled at Skåne University Hospital in Lund, Sweden. The trial is investigator-initiated and non-commercial.

POPULATION AND INTERVENTION Adults (18 years of age or older) in need of a subclavian CVC for any reason and able to give written informed consent will be included in the study provided no exclusion criteria is fulfilled.

OUTCOMES Primary outcome will be number of CVC insertions with >1 skin puncture. Secondary outcomes include comparison between the two groups regarding 1) the frequency of mechanical complications, 2) proportion of the insertion-time when the needle is visible on the ultrasound (US) screen, 3) time to successful vessel punction, 4) the number of needle redirections during the insertion, 5) number of failed catheterisations, 6) Feasibility of the needle guide evaluated with a questionair to the operators at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients in need of a central venous catheter .
* Clinical indication for the subclavian route which includes expected time of use >5 days.
* Signed informed consent.

Exclusion Criteria:

* Patient is deemed unsuitable for cannulation of the subclavian vein, based on a pre-procedural US examination by the operator, or due to unacceptable patient risk in case of mechanical complication (e.g., severe respiratory failure).

Ages: 18 Years to 105 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2022-11-08 (Actual); Primary Completion 2025-09-16 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
Number of subclavian catheter insertions with >1 skin puncture | During the central venous catheterization, up to 3 hours after inclusion
  Number of subclavian catheter insertions with >1 skin puncture

SECONDARY OUTCOMES:
The frequency of mechanical complications | 24 hours after the completion of the central venous catheterization
  Mechanical complication include: 1) Bleeding World Health Organization (WHO)-grade 2-4. 2) Pneumothorax visible on post-procedural Xray. 3) Permanent nerve injury. 4) Arrhythmia WHO-grade 3 and 4. 5) Arterial catheterization
Needle visibility | During the central venous catheterization, up to 4 hours after inclusion
  Proportion of the insertion-time when the needle is visible on the ultrasound screen
Time to successful vessel puncture | During the central venous catheterization, up to 4 hours after inclusion
  Time to successful vessel puncture
The number of needle redirections | During the central venous catheterization, up to 4 hours after inclusion
  The number of needle redirections during the insertion
The number of failed catheterizations | During the central venous catheterization, up to 4 hours after inclusion
  The number of failed catheterizations in the attempted subclavian vein
Feasibility of the needle guide | Through the study period, anticipated 3 years
  Feasibility of the needle guide by means of a questionnaire at the end of the study period.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Kander, Assoc. Prof., Principal Investigator — Region Skåne and Lund University
Locations (1):
- Intensive and Perioperative Care. Skåne University Hospital. Lund, Lund, Skåne County, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this study, will be made available on reasonable request and after deidentification.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data will be available beginning 3 months and ending 5 years following article publication.
Access Criteria: Access will be given to researchers who provide a methodologically sound proposal. Proposals should be directed to the research group Clinical Research in Anaesthesia and Intensive Care Medicine, C/O Thomas Kander, Dept. of Clinical Sciences, Lund, Lund University, Sweden. To gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- [Derived] Naddi L, Borgquist O, Adrian M, Bark BP, Kander T. Ultrasound-guided subclavian vein catheterisation with a needle guide (ELUSIVE): protocol for a randomised controlled study. BMJ Open. 2023 Dec 19;13(12):e080515. doi: 10.1136/bmjopen-2023-080515. PMID 38114277